CLINICAL TRIAL: NCT04300244
Title: Nivolumab and Ipilimumab +/- UV1 Vaccination as Second Line Treatment in Patients With Malignant Mesothelioma (the NIPU-study)
Brief Title: Nivolumab and Ipilimumab +/- UV1 Vaccination as Second Line Treatment in Patients With Malignant Mesothelioma
Acronym: NIPU
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Åslaug Helland (Other)
Collaborators: Oslo University Hospital (Other); Ultimovacs ASA (Industry); Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor-Investigator, Åslaug Helland, MD, Prof, PhD, Ullevaal University Hospital
Organization: Oslo University Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CA209-7H4 NIPU
Record Dates: First submitted 2020-02-19; First posted 2020-03-09 (Actual); Last update posted 2024-02-29 (Actual); Status verified 2024-02

CONDITIONS: Cancer; Cancer, Lung; Cancer of Lung; Mesothelioma; Mesothelioma; Lung; Mesothelioma; Pleura; Mesotheliomas Pleural
MeSH Terms: conditions — Neoplasms; Lung Neoplasms; Mesothelioma; Mesothelioma, Malignant | interventions — UV1 vaccine; sargramostim; Ipilimumab; Nivolumab

STUDY DESIGN:
Intervention Model Description: randomized, multi-center, open-label, proof of concept study comparing the efficacy and safety of nivolumab and ipilimumab with or without UV1 in patients with inoperable malignant pleural mesothelioma after first-line platinum-based chemotherapy.
Masking Description: Open label
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Arm A (Experimental): Ipilimumab and nivolumab + UV1
  Interventions: Biological: UV1 vaccine + leukine; Biological: ipilimumab; Biological: nivolumab
- Arm B (Active Comparator): Ipilimumab and nivolumab
  Interventions: Biological: ipilimumab; Biological: nivolumab

INTERVENTIONS:
Biological: UV1 vaccine + leukine — The mode of action of UV1 is to activate the immune system to induce T cells directed against telomerase (hTERT). UV1 vaccination amplifies the pool of hTERT specific tumor-reactive T cells from the naive repertoire and has the potential to increase the breadth and diversity of the tumor-reactive T cell response (epitope spreading). Vaccination with UV1 can thus provide the basis for increased efficacy of checkpoint inhibition therapy, by augmenting the pool of tumor specific T cells in patients with limited or insufficient numbers of T cell clones spontaneously primed by tumor antigens. Reciprocally, the efficacy of UV1 vaccination may be enhanced in combination with checkpoint inhibitors, since the clonal expansion and effector activity of UV1 induced T cells will otherwise be restricted by intrinsic immune regulatory and tumor induced suppressor mechanisms.
  Arms: Arm A
Biological: ipilimumab — The responses to ipilimumab and nivolumab combination therapy seen in MPM is encouraging.
  Other Names: Yervoy
Biological: nivolumab — The responses to ipilimumab and nivolumab combination therapy seen in MPM is encouraging.
  Other Names: Opdivo

SUMMARY:
The objective of the study is to induce a meaningful progression-free survival benefit in patients with Malign Pleural Mesothelioma (MPM) after progression on first line standard platinum doublet chemotherapy, by treating with nivolumab and ipilimumab with or without UV1 vaccine.

DETAILED DESCRIPTION:
Several studies have investigated the use of checkpoint inhibition in Malign Pleural Mesothelioma (MPM). Most of them are small studies investigating the efficacy of single-agent immunotherapy in few patients. Given that the combination of anti-PD-1 or anti-PD-L1 therapy with CTLA-4 has been shown in other cancers to enhance treatment effect, combined checkpoint inhibitor treatment has also been investigated in patients with MPM. Although these results are encouraging, the response rates seen are moderate compared to what has been documented for the combination of checkpoint inhibitors in other cancer indications. An approach to further enhance the PFS and response rate in MPM may be to use a vaccine aiming to activate an immune response directed against tumor-related antigens, and to combine the vaccine with checkpoint inhibitors. The proposed study will evaluate the use of the therapeutic cancer vaccine UV1 in combination with nivolumab and ipilimumab after progression on standard first-line chemotherapy in patients with malignant pleural mesothelioma.

The objective of the study is to induce a meaningful progression-free survival benefit in patients with MPM after progression on first line standard platinum doublet chemotherapy, by treating with nivolumab and ipilimumab with or without UV1.

The primary end-point (PFS) is expected to be analyzed in 2023.

ELIGIBILITY:
Inclusion Criteria:

* Histologically and/or cytologically confirmed malignant pleural mesothelioma.
* Unresectable disease
* Measurable disease, defined as at least 1 lesion (measurable) that can be accurately assessed at baseline by computed tomography (CT) or magnetic resonance imaging (MRI) and is suitable for repeated assessment (modified RECIST).
* Available unstained archived tumor tissue sample in sufficient quantity to allow for analyses. At least fifteen unstained slides or a tumor block (preferred). NOTE: A fine needle aspiration sample is not sufficient to make the patient eligible for enrollment. Given the complexity of mesothelioma pathological diagnosis , it is expected that they will have a core needle biopsy or surgical tumor biopsy as part of their initial diagnostic work up.
* Age ≥ 18 years.
* Eastern Cooperative Oncology Group (ECOG) performance status of 0 - 1.
* Willing to provide archived tumor tissue and blood samples for research.
* Adequate organ function as defined below

  1. Haemoglobin ≥ 9.0 g/dL
  2. Absolute neutrophil count (ANC) 1.5 (or 1.0) x (> 1500 per mm3)
  3. Platelet count ≥100 (or 75) x 109/L (>75,000 per mm3)
  4. Serum bilirubin ≤1.5 x institutional upper limit of normal (ULN).
  5. AST (SGOT)/ALT (SGPT) ≤2.5 x institutional upper limit of normal unless liver metastases are present, in which case it must be ≤5x ULN
  6. Measured creatinine clearance (CL)

     1. >40 mL/min
     2. Calculated creatinine CL>40 mL/min (Cockcroft-Gault formula)
     3. 24-hour urinecollection for determination of CL
* Males: Creatinine CL (mL/min) =Weight (kg) x (140 - Age) 72 x serum creatinine (mg/dL)
* Females:Creatinine CL (mL/min)=Weight (kg) x (140 - Age)x0.85 72 x serum creatinine (mg/dL)
* Previously treated with at least one line of platinum -pemetrexed

Exclusion Criteria:

* Disease suitable for curative surgery
* Previous treatment with a PD-1 or PD-L1 inhibitor, including nivolumab or any other agent targeting immune checkpoints.
* Non-pleural mesothelioma e.g. mesothelioma arising in peritoneum, tunica vaginalis or any serosal surface other than the pleura.
* Active second malignancy other than non-melanoma skin cancer or cervical carcinoma in situ.
* Symptomatic or uncontrolled brain metastases requiring concurrent treatment, inclusive of but not limited to surgery, radiation and/or corticosteroids (prednisone >10 mg or equivalent). Surgery, radiation and/or corticosteroids (any dose >10 mg prednisone equivalent) must have been completed ≥ 2 weeks prior to registration.
* Uncontrolled seizures.
* Current or prior use of immunosuppressive medication within 28 days before the first dose of nivolumab, with the exceptions of intranasal and inhaled corticosteroids or systemic corticosteroids at physiological doses, which are not to exceed 10 mg/day of prednisone, or an equivalent corticosteroid. Standard steroid premedication given prior to chemotherapy or as prophylaxis for imaging contrast allergy should not be counted for this criterion.
* Active or prior documented autoimmune or inflammatory disorders (including inflammatory bowel disease, diverticulitis with the exception of diverticulosis, celiac disease, irritable bowel disease; Wegner syndrome) within the past 2 years. Subjects with vitiligo, alopecia, Grave's disease, or psoriasis not requiring systemic treatment (within the past 3 years) are not excluded.
* History of primary immunodeficiency.
* History of allogeneic organ transplant.
* Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, uncontrolled hypertension, unstable angina pectoris, cardiac arrhythmia, active peptic ulcer disease or gastritis, active bleeding diatheses including any subject known to have psychiatric illness/social situations that would limit compliance with study requirements or compromise the ability of the subject to give written informed consent.
* Active infection including tuberculosis (clinical evaluation including: physical examination findings, radiographic findings, positive PPD test, etc.), hepatitis B (known positive HBV surface antigen [HBsAg] result), hepatitis C, or human immunodeficiency virus (positive HIV 1/2 antibodies as defined by a positive ELISA test). Patients with a past or resolved HBV infection (defined as the presence of hepatitis B core antibody [anti-HBc] and absence of HBsAg) are eligible. Patients positive for hepatitis C (HCV) antibody are eligible only if polymerase chain reaction is negative for HCV RNA. HIV testing is not required in the absence of clinical suspicion.
* Known history of leptomeningeal carcinomatosis.
* Pregnant or lactating women
* Live attenuated vaccination within 30 days prior to study entry or within 30 days of receiving nivolumab.
* Any condition that, in the opinion of the investigator, would interfere with the evaluation of study treatment or interpretation of patient safety or study results.
* History of allergy or hypersensitivity to any of the active substances or excipients in the study drug.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 118 (Estimated)
Dates: Start 2020-05-04 (Actual); Primary Completion 2025-03-15 (Estimated); Study Completion 2027-03-15 (Estimated)

PRIMARY OUTCOMES:
Evaluation of efficacy of ipilimumab and nivolumab With or without UV1 vaccine in patients With inoperable malignant pleural mesothelioma progressing after first-line platinum-based chemotherapy. | Monitoring for change in imaging evalated tumor lesions indicating progression throughout the trial until 5 years of follow-up has past.
  Progression-free survival (PFS) per Modified Response Evaluation Criteria in Solid Tumors (RECIST) as determined by blinded independent central review (BICR) assessed by radiologic assessments

SECONDARY OUTCOMES:
Response evaluation | Throughout the trial. Radiological assessments every 6th week during the first year, every 12th week for the next 5 years.
  Comparison of response rate according to Response Evaluation Criteria in Solid Tumors, version 1.1 (Modified RECIST), in patients who receive nivolumab and ipilimumab with patients who receive nivolumab and ipilimumab in combination with UV1.
Evaluation of patient reported outcomes (PRO) | every other week for the first 12 weeks, every 6th week thereafter
  To evaluate changes from baseline in patient-reported outcomes (PROs) in patients who receive nivolumab and ipilimumab compared to patients who receive nivolumab and ipilimumab in combination with UV1.
Evaluation of Adverse Events and discontinuation rate of patients | Continuously, and until 90 days after discontinuation of study treatment.
  To determine the safety and tolerability of patients receiving ipilimumab and nivolumab With or without UV1 vaccination by monitoring AEs and study drug discontinuation due to AEs.
  tolerability in patients who receive nivolumab and ipilimumab compared to patients who receive nivolumab and ipilimumab in combination with UV1, measured by adverse events (AE) and study drug discontinuations due to AEs.

OTHER OUTCOMES:
Assessment of repertoire of TCR specificities induced by UV1 vaccination | blood samples collected at screening, week 6, week 12 and week 18/19.
  Generating TCR repertoire data and comparing differences pre- and post treatment between the two treatment arms
Investigate whether there is a correlation between baseline tumor mutational burden (TMB) and response to therapy | In tissue collected at screening, week 5/6, and study completion, at most 2 years.
  Characterization of TMB pre- and post-treatment by DNA analyses of tumor and normal tissue to identify tumor-specific somatic mutations, and comparing results to clinical outcome data.
investigate whether there is a difference in the immune cell infiltrate in the tumor pre- and post treatment With UV1 and check point inhibition. | In tissue collected at screening, week 5/6, and study completion, at most 2 years.
  By characterizing qualitative and quantitative differences in markers of immune activation within tumor samples pre and post therapy by immunohistochemistry.
Investigate whether UV1 vaccination induces hTERT-specific T cells in the blood of patients treated. | blood samples collected at pre-defined evaluation points throughout study completion, at most 2 years.
  By detection of vaccine-specific T cells in PBMC harvested from patients by T cell proliferation assays
Investigate whether DTH response correlates With detection of a vaccine-specific T cell response in blood | blood samples collected atat pre-defined evaluation points throughout study completion, at most 2 years.
  The trial will compare DTH measurements With vaccine-specific T-cell response in blood.
Investigate whether there is a correlation between the microenvironment in feces and treatment response. | blood samples collected at at pre-defined evaluation points throughout study completion, at most 2 years.
  Stool samples will be collected and data on microbial gut composition for each patient will be correlated With treatment outcome.

CONTACTS AND LOCATIONS:
Overall Officials: Åslaug Helland, Prof, MD, Principal Investigator — Oslo University Hospital
Locations (7):
- University of Western Australia, Perth, Australia
- Denmark (2):
  - Aalborg University Hospital, Aalborg
  - Copenhagen University Hospital, Copenhagen
- Oslo University Hospital, Oslo, Norway
- Vall d'Hebron institute of oncology, Barcelona, Spain
- Sweden (2):
  - University Hospital of Skåne, Lund
  - Karolinska, Stockholm

REFERENCES:
- [Derived] Thunold S, Hernes E, Farooqi S, Ojlert AK, Francis RJ, Nowak AK, Szejniuk WM, Nielsen SS, Cedres S, Perdigo MS, Sorensen JB, Meltzer C, Mikalsen LTG, Helland A, Malinen E, Haakensen VD. Outcome prediction based on [18F]FDG PET/CT in patients with pleural mesothelioma treated with ipilimumab and nivolumab +/- UV1 telomerase vaccine. Eur J Nucl Med Mol Imaging. 2025 Jan;52(2):693-707. doi: 10.1007/s00259-024-06853-0. Epub 2024 Aug 12. PMID 39133306
- [Derived] Haakensen VD, Nowak AK, Ellingsen EB, Farooqi SJ, Bjaanaes MM, Horndalsveen H, Mcculloch T, Grundberg O, Cedres SM, Helland A. NIPU: a randomised, open-label, phase II study evaluating nivolumab and ipilimumab combined with UV1 vaccination as second line treatment in patients with malignant mesothelioma. J Transl Med. 2021 May 31;19(1):232. doi: 10.1186/s12967-021-02905-3. PMID 34059094